CLINICAL TRIAL: NCT06095271
Title: A Multicenter, Randomized Pragmatic Platform Trial Embedded Within the Swiss Multiple Sclerosis Cohort (SMSC) on Neurofilament Light Chain Monitoring Added to Usual Care to Inform Personalized Treatment Decisions in Multiple Sclerosis
Brief Title: MultiSCRIPT-Cycle 1: Personalized Medicine in Multiple Sclerosis - Pragmatic Platform Trial Embedded Within the SMSC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MultiSCRIPT-Cycle 1
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sNfL monitoring (Experimental): 6-monthly blood draw to measure sNfL
  Interventions: Diagnostic Test: serum Neurofilament Filament Light chain (sNfL) monitoring
- Usual care (No Intervention): SMSC usual care

INTERVENTIONS:
Diagnostic Test: serum Neurofilament Filament Light chain (sNfL) monitoring — the intervention consist of a blood draw and providing the sNfL information to the treating physician
  Arms: sNfL monitoring

SUMMARY:
This is a randomized pragmatic clinical trial fully embedded in the Swiss Multiple Sclerosis Cohort to assess whether sNfL biomarker monitoring improves patient-relevant outcomes and care of patients with relapsing-remitting (RR)MS by either increasing the proportion of patients with no evidence of disease activity (EDA) or by improving patients' health-related quality of life.

DETAILED DESCRIPTION:
The course of multiple sclerosis (MS) is highly heterogenous with a large variability in symptoms, severity and response to treatment. A large majority of persons with MS are treated with disease modifying therapies (DMTs). DMTs can dramatically reduce even almost suppress relapses and occurrence of new lesions in magnetic resonance imaging (MRI) by weakening the immune system but which in turn may cause side effects such as opportunistic infections with prolonged treatment duration and intensity of the immunosuppression.

A more personalized approach to MS therapy is urgently needed to treat patients as little as possible but as much as necessary and at the right time. Such tailored strategies cannot be made without detailed information on treatment response and disease activity. Levels sNfL, which is released in the blood following neuroaxonal damage, has been shown to be associated with future MS disease activity, disability worsening, MRI activity and treatment response. sNfL might therefore be helpful for a patient-tailored treatment adaptation (e.g., escalation or de-escalation) ensuring disease stability, fewer adverse events and better quality of life. While sNfL is increasingly used as a marker of treatment response, its use in routine care is not yet widely established.

The SMSC is an observational study across 8 Swiss leading MS centers including >1600 participants with MS with a median follow-up of >5.7 years. The MultiSCRIPT project aims to use this real-world data infrastructure to systematically evaluate patient-relevant benefits resulting from innovations in MS patient care.

MultiSCRIPT goes beyond a unique trial but aims to be a sustainable learning system in which accumulating data from successive pragmatic randomized trials (i.e., learning cycles) enable the continuous generation of new hypotheses on how treatment and care strategies can be further personalized to treat patients as little as possible but as much as necessary at the right time. By being nested within the already existing and ongoing SMSC, this research infrastructure embedded in clinical care offers an unique opportunity to efficiently conduct a nationwide real-life evaluation of new care strategies, at low costs, and fostering evaluation and direct translation of effective innovations into usual care to improve patient outcome and quality of life. MultiSCRIPT-Cycle 1 is the first learning cycle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RRMS according to the most recent McDonald criteria (2017) for at least one year
* Have already consented to take part in the SMSC
* Age 18 years old or older
* Able and willing to consent

Exclusion Criteria:

* Inclusion or planned inclusion in another clinical trial that determines the drug therapy for MS for the purpose of research as these patients are most likely not following the SMSC usual care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
EDA3 (evidence of disease activity) | 24-months
  number of participant with a relapse or disability worsening (measured by Expanded Disability Status Scale (EDSS)) or disease activity on MRI imaging (new/enlarging T2 weighted lesions or T1 weighted contrast enhancing lesion on cranial or spinal cord MRI)
Multiple Sclerosis Quality of Life (MSQOL)-54 Instrument | 24-months
  The summary scores are the physical health composite summary and the mental health composite summary. A higher score indicates improved quality of life

SECONDARY OUTCOMES:
Multiple Sclerosis Quality of Life (MSQOL)-54 Instrument | 12-months
  The summary scores are the physical health composite summary and the mental health composite summary. A higher score indicates improved quality of life
EDA3 (evidence of disease activity) | 12-months
  number of participant with a relapse or disability worsening (measured by Expanded Disability Status Scale (EDSS)) or disease activity on MRI imaging (new/enlarging T2 weighted lesions or T1 weighted contrast enhancing lesion on cranial or spinal cord MRI)
EQ-5D-5L | 12- and 24-months
  The EQ-5D-5L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and includes an overall visual analog scale
Short form 36 (SF-36) | 12- and 24-months
  contained in the MSQoL-54 questionnaire. The lower the score the more disability.
relapses | 12- and 24-months
  according to McDonald criteria
disability worsening | 12- and 24-months
  measured by Expanded Disability Status Scale (EDSS). The EDSS ranges from 0 to 10. The greater the level of disability, the higher is the score.
New/enlarging T2w lesions | 12- and 24-months
  MRI imaging
T1w contrast enhancing lesions | 12- and 24-months
  MRI imaging
Amount of immunosuppressive/immunomodulatory drug treatment | 12- and 24-months

OTHER OUTCOMES:
Serious adverse events related to blood draw | up to 42-months
Mortality | up to 42-months
Adverse events related to immunosuppression | up to 42-months
Occurrence of relapses in patients previously stable | up to 42-months
  according to McDonald criteria
Disability worsening in patients previously stable | up to 42-months
  measured by Expanded Disability Status Scale (EDSS). The EDSS ranges from 0 to 10. The greater the level of disability, the higher is the score.

CONTACTS AND LOCATIONS:
Overall Officials: Özgür Yaldizli, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (8):
- Switzerland (8):
  - University Hospital Basel, Basel, Canton of Basel-City
  - Kantonsspital Aarau, Aarau
  - Inselspital Bern, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Ospedale Regionale di Lugano, sede Civico, Lugano
  - Kantonsspital St.Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich

REFERENCES:
- [Derived] Janiaud P, Zecca C, Salmen A, Benkert P, Schadelin S, Orleth A, Demuth L, Maceski AM, Granziera C, Oechtering J, Leppert D, Derfuss T, Achtnichts L, Findling O, Roth P, Lalive P, Uginet M, Muller S, Pot C, Hoepner R, Disanto G, Gobbi C, Rooshenas L, Schwenkglenks M, Lambiris MJ, Kappos L, Kuhle J, Yaldizli O, Hemkens LG. MultiSCRIPT-Cycle 1-a pragmatic trial embedded within the Swiss Multiple Sclerosis Cohort (SMSC) on neurofilament light chain monitoring to inform personalized treatment decisions in multiple sclerosis: a study protocol for a randomized clinical trial. Trials. 2024 Sep 11;25(1):607. doi: 10.1186/s13063-024-08454-6. PMID 39261900